CLINICAL TRIAL: NCT03638440
Title: Real World Observational Study of Naloxegol for Patients With Cancer Pain Diagnosed With Opioid Induced Constipation.
Brief Title: Real World Observational Study of Naloxegol for Patients With Cancer Pain Diagnosed With OIC.
Acronym: NACASY
Status: Completed | Type: Observational
Sponsor: Kyowa Kirin Pharmaceutical Development Ltd (Industry)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: NACASY
Record Dates: First submitted 2018-08-07; First posted 2018-08-20 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Opioid Induced Constipation
Keywords: Opioid Induced Constipation; Naloxegol; Peripherally Acting Mu-Opioids Receptor Antagonist (PAMORA)
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Naloxegol — Naloxegol is a PEGylated derivative of the μ-opioid receptor antagonist naloxone
  Other Names: Moventig

SUMMARY:
This is a single-arm, open label, multinational, multicentre, prospective, real world observational study of Naloxegol in adult subjects with Opioid Induced Constipation (OIC) in patients receiving Naloxegol in routine clinical practice. Subjects who are receiving Naloxegol (prescribed by their physician according to the SmPC, which recommends that all currently used maintenance laxative therapy should be halted) during the enrolment period may be eligible for enrolment into the study.

DETAILED DESCRIPTION:
The objective of this study is to assess the safety and efficacy of Naloxegol in a real world setting in cancer patients.

The primary safety end point is the incidence of adverse events leading to study discontinuation.

The primary efficacy end point is the response rate assessed in the 4 week observation period. Response is defined as three or more bowel movements (without the use of rescue laxative treatment in the previous 24 hours) per week and an increase of one or more bowel movements over baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient who is receiving treatment with opioids for at least 4 weeks, and is expected to remain on opioids for duration of study
* Patient with opioid-induced constipation
* Patient in whom the clinician plans treatment with Naloxegol according to routine clinical practice (Naloxegol SmPC recommends that all currently used maintenance laxative therapy should be halted)
* Signing of the informed consent

Exclusion Criteria:

- Patients with colorectal cancer

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will involve 315 patients (out-patients or in-patients) with Opioid Induced Constipation (OIC) from 32 European hospitals.
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
To assess the safety and efficacy of Naloxegol in a real world setting in cancer patients. | 4 week treatment period
  Response rate

SECONDARY OUTCOMES:
Proportion of patients that have a BFI score change of ≥12 points at the end of the study treatment | 4 week observation period
  Bowel Function Index (BFI) score change of ≥12 points
Proportion of patients that have a BFI score <30 at the end of the study (patients adequately treated). | 4 week observation period
  Bowel Function Index (BFI) score <30
Time to the first post-dose bowel movement | 4 week observation period
  Time to first post-dose bowel movement
Change in stool consistency | 4 week observation period
  Bristol stool scale (BSS)
Change in Patient Assessment of Constipation (PAC-QOL) | 4 week observation period
  Quality of Life Questionnaire
Incidence of overall adverse events, including SAEs | 4 week observation period
  Adverse Events, including SAEs
Analgesic treatment interruptions/dose adjustments | 4 week observation period
  Dose adjustments
Naloxegol treatment interruptions/dose adjustments | 4 week observation period
  Dose adjustments
Patient satisfaction (PGI-I) | 4 week observation period
  Patient Global Impression of Improvement (PGI-I)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, MD, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust; Jan Tack, MD, Principal Investigator — University Hospital KU Leuven
Locations (10):
- Aalborg University Hospital, Aalborg, Denmark
- Tampere University Hospital, Tampere, Finland
- Paul Papin à Angers et site René Gauducheau, Nantes, France
- Lubecker Onkologische, Lübeck, Germany
- Areteion Hospital, Athens, Greece
- AORN dei Colli, Napoli, Italy
- Rijnstate hospital, Arnhem, Netherlands
- ICO-Hospitalet, Barcelona, Spain
- Skane University Hospital, Lund, Sweden
- Royal Surrey County Hospital, Guildford, Surrey, United Kingdom